CLINICAL TRIAL: NCT04816253
Title: Methylprednisolone and Hyaluronic Acid Versus Each Agent Alone to Control Post-extraction Complications of Impacted Mandibular Third Molar
Brief Title: Controlling Post-extraction Complications of Impacted Mandibular Third Molar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Alaa Altaweel, Associate professor, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Extraction healing
Record Dates: First submitted 2021-03-23; First posted 2021-03-25 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Preventing Postextraction Complication
MeSH Terms: interventions — Saline Solution; Hyaluronic Acid; Methylprednisolone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Normal saline (Placebo Comparator): Normal saline irrigation after extraction and No drug placed in tooth socket
  Interventions: Drug: Normal saline
- Gengigel (Active Comparator): Gengigel (Hyaluronic acid) placed after extraction
  Interventions: Drug: Hyaluronic acid
- Methylprednisolone (Active Comparator): Methylprednisolone will be given intravenous to a patient half an hour before the surgery
  Interventions: Drug: Methylprednisolone
- Methylprednisolone and Gengigel (Active Comparator): Methylprednisolone will be given intravenous to a patient half an hour before the surgery and Gengigel (Hyaluronic acid) placed after extraction
  Interventions: Drug: Methylprednisolone and Hyaluronic acid

INTERVENTIONS:
Drug: Normal saline — Normal saline irrigation and No other drug placed after extraction
  Arms: Normal saline
Drug: Hyaluronic acid — Immediately after removal of impacted tooth (hyaluronic acid) placed in extraction socket
  Other Names: Gengigel
  Arms: Gengigel
Drug: Methylprednisolone — Methylprednsolone will be injected half an hour preoperatively
  Arms: Methylprednisolone
Drug: Methylprednisolone and Hyaluronic acid — Methylprednisolone will be injected half an hour preoperatively and Immediately after removal of impacted tooth (hyaluronic acid) placed in extraction socket
  Arms: Methylprednisolone and Gengigel

SUMMARY:
Impacted mandibular 3rd molar will be extracted in all patients, then patients will be divided, according to material placed in extraction socket into 3 groups: control, hyaluronic acid and honey. Then post extraction complications will be evaluated

DETAILED DESCRIPTION:
Impacted Mandibular third molar will be extracted under local anesthesia Through standard surgical flap elevation, after extraction and wound irrigation a material facilitate healing will be placed. According to material will be placed patients will be divide into 3 group: control ( no material, second group hyaluronic acid, third group ( honey).. then wound will be closed. Postoperative pain ( through visual analog scale) , edema, total dose of analgesic, mandibular movement (interincisal distance in mm) will be evaluated preoperative, 1,2,3,7, and 10 day after extraction

ELIGIBILITY:
Inclusion Criteria:

* healthy patients
* patient has impacted 3rd molar

Exclusion Criteria:

* medically compromised patients Heavy smoking patients

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2021-06-20 (Actual)

PRIMARY OUTCOMES:
Interincisal distance | Baseline (Preoperative)
  Measuring distance between upper lower anterior teeth in mm
Interincisal distance | 1 day postoperative
  Measuring distance between upper lower anterior teeth in mm
Interincisal distance | 2nd day postoperative
  Measuring distance between upper lower anterior teeth in mm
Interincisal distance | 3rd day postoperative
  Measuring distance between upper lower anterior teeth in mm
Interincisal distance | 7th day postoperative
  Measuring distance between upper lower anterior teeth in mm
Assessment of pain using Visual analog scale | Baseline (Preoperative)
  Patient asked to describe pain intensity subjectively on visual analog scale where 0 mean no pain while 10 mean sever pain
Assessment of pain using Visual analog scale | 1st day
  Patient asked to describe pain intensity subjectively on visual analog scale where 0 mean no pain while 10 mean sever pain
Assessment of pain using Visual analog scale | 2nd day
  Patient asked to describe pain intensity subjectively on visual analog scale where 0 mean no pain while 10 mean sever pain
Assessment of pain using Visual analog scale | 3rd day
  Patient asked to describe pain intensity subjectively on visual analog scale where 0 mean no pain while 10 mean sever pain
Assessment of pain using Visual analog scale | 7th day
  Patient asked to describe pain intensity subjectively on visual analog scale where 0 mean no pain while 10 mean sever pain
Total amount of analgesic | 1st day postoperative
  Total amount of analgesic Will be calculated
Total amount of analgesic | 2nd day postoperative
  Total amount of analgesic Will be calculated
Total amount of analgesic | 3rd day postoperative
  Total amount of analgesic Will be calculated
Total amount of analgesic | 7th day postoperative
  Total amount of analgesic Will be calculated
Size of edema will be assessed from finial angle and Travis of ear to mental ala of Nes and mouth angle | Baseline
  Edema measured from gonial angle and Tragus to mental, angle of mouth, ala of nose, and lateral canthus of eye respectively
Size of edema will be assessed from finial angle and Travis of ear to mental ala of Nes and mouth angle | 1st day postoperative
  Edema measured from gonial angle and Tragus to mental, angle of mouth, ala of nose, and lateral canthus of eye respectively
Size of edema will be assessed from finial angle and Travis of ear to mental ala of Nes and mouth angle | 2nd day postoperative
  Edema measured from gonial angle and Tragus to mental, angle of mouth, ala of nose, and lateral canthus of eye respectively
Size of edema will be assessed from finial angle and Travis of ear to mental ala of Nes and mouth angle | 3rd day postoperative
  Edema measured from gonial angle and Tragus to mental, angle of mouth, ala of nose, and lateral canthus of eye respectively
Size of edema will be assessed from finial angle and Travis of ear to mental ala of Nes and mouth angle | 7th day postoperative
  Edema measured from gonial angle and Tragus to mental, angle of mouth, ala of nose, and lateral canthus of eye respectively

CONTACTS AND LOCATIONS:
Locations (1):
- Vision college, Jeddah, Saudi Arabia